CLINICAL TRIAL: NCT00263770
Title: A Randomized, Controlled Treatment Trial of Soft Palatal Implants and Positive Airway Pressure in Mild to Moderate Obstructive Sleep Apnea and Snoring
Brief Title: Treatment Study of Soft Palatal Implants in Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Medtronic Xomed, Inc. (Industry); ResMed Foundation (Other)
Responsible Party: Sean M Caples, D.O, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1646-05; 5591559902
Record Dates: First submitted 2005-12-07; First posted 2005-12-09 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Positive airway pressure (PAP) (Other): which is air delivered by a mask worn over the nose during sleep
  Interventions: Other: Positive airway pressure (PAP)
- outpatient surgical procedure (Active Comparator): where small fabric rods are inserted into the soft palate (the fleshy portion of the roof of the mouth) to stiffen the tissues.
  Interventions: Device: soft palate implant
- Sham surgery (Sham Comparator): an outpatient surgical procedure identical to #2 except that no rods are inserted into the soft palate.
  Interventions: Device: soft palate implant

INTERVENTIONS:
Device: soft palate implant
  Arms: Sham surgery; outpatient surgical procedure
Other: Positive airway pressure (PAP) — which is air delivered by a mask worn over the nose during sleep
  Arms: Positive airway pressure (PAP)

SUMMARY:
The purpose of the study is to compare the effectiveness of soft palatal implants with placebo and continuous positive airway pressure treatment in obstructive sleep apnea.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA), frequently associated with disruptive snoring, is a prevalent disorder which is increasingly recognized by health care providers and lay people alike as an important factor in impaired daytime executive function as well as cardiovascular disease risk. Along with an increase in its recognition and diagnosis have come a growing pool of patients with milder disease and the associated challenge of ideal management. Positive airway pressure (PAP) is well established as the mainstay of treatment for OSA since it is effective at reversing daytime neurocognitive sequelae and may be a useful adjunct to therapy in those with cardiovascular disease coexisting with OSA. In patients with mild OSA, however, the response to PAP therapy appears muted, which is related in part to poor adherence to treatment. In response, a number of alternative treatments have evolved. The most recent innovation is soft palatal implants, which, in non-randomized, uncontrolled studies have demonstrated reasonable efficacy in the treatment of snoring and mild to moderate OSA. How the implants compare with standard therapy and their effect on cardiovascular variables are unknown. Because of the ease and rapidity with which this system is implanted, and because treatment effect is independent of patient compliance, there is high potential for widespread use in patients with milder OSA. We therefore are conducting a randomized, placebo-controlled clinical trial to compare the impact of palatal implants with PAP on sleep disordered breathing, daytime symptoms and blood pressure, as well as patient / bed partner acceptance.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age >18 yrs
2. AHI 5-30
3. Tonsil size <50% of airway
4. No anatomically fixed nasal stenosis
5. BMI = 32 kg/m2 EXCLUSION CRITERIA

1. The presence of a concomitant untreated primary sleep disorder (restless legs syndrome, narcolepsy, idiopathic hypersomnia) 2. Severe daytime sleepiness (history of sleep-related motor vehicle or occupational accident) 3. Moderate to severe pulmonary disease (FEV1 <50% pred) 4. Neurologic impairment (h/o CVA, TIA, neuromuscular disease, diaphragmatic paralysis) 5. Significant cardiac disease (LVEF<50%, moderate to severe valvular disease) 6. Uncontrolled hypertension >180/110 7. Renal disease (Scr > 2.5) 8. Allergy to local anesthetics used for implantation procedure. 9. Pregnant or nursing women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
apnea-hypopnea index | 90 days

SECONDARY OUTCOMES:
sleepiness | 90 days
quality of life | 90 days
ambulatory blood pressure | 90 days
snoring | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Sean M. Caples, D.O., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States